CLINICAL TRIAL: NCT00823446
Title: A Feasibility, Double Blind, Randomized, Controlled Clinical Study to Evaluate the Safety of Topically Applied Revera vs. Control in Subjects With Venous Leg Ulcers.
Brief Title: Feasibility Study to Evaluate the Safety of Topically Applied Revera in Subjects With Venous Leg Ulcers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Revalesio Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RC 03.1.1.HS1
Record Dates: First submitted 2009-01-13; First posted 2009-01-15 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Venous Stasis Ulcers
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Revera Wound Care (Experimental)
  Interventions: Device: Revera Wound Care
- Normal Saline (Placebo Comparator)
  Interventions: Device: Normal Saline

INTERVENTIONS:
Device: Revera Wound Care — Revalesio Part Number MDW0060
  Arms: Revera Wound Care
Device: Normal Saline — Sodium Chloride for Irrigation
  Arms: Normal Saline

SUMMARY:
The purpose of this study is to perform a preliminary evaluation of the safety of Revera Wound Care when topically applied to venous leg ulcers for 8 weeks of treatment.

DETAILED DESCRIPTION:
The purpose of this study is to perform a preliminary evaluation of the safety of Revera Wound Care when topically applied to venous leg ulcers for 8 weeks of treatment.

This evaluation will be done through tabulations of adverse events (AE), review of complete blood counts (CBC) with differential and platelet, and measuring wound healing rate.

The secondary purpose of the study is a preliminary evaluation of an increase in the healing rate of venous leg ulcers treated with Revera Wound Care.

This evaluation will be done through measuring wound healing rate (which is also being used to evaluate safety) and complete wound healing.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Diagnosis of non-healing venous leg ulcer by the following criteria:

  * dependent peripheral edema, dermatitis, hyperpigmentation.
  * an ankle to arm arterial pressure ratio > 0.7 as measured by arterial Doppler.
* Venous Stasis Ulcer is ≥ 2 cm² in size.
* If female subject of reproductive age, have had a negative pregnancy test within one week of study entry and are using adequate birth control.

Exclusion Criteria:

* Subject known to be allergic to Aquacel dressing or components.
* Peripheral arterial insufficiency (as determined by Doppler ABI), uncontrolled congestive heart failure (CHF), vasculitis, uncontrolled diabetes mellitus.
* Severe contact dermatitis (allowable if it does not interfere with application of the dressings).
* Concomitantly receiving systemic corticosteroids in doses exceeding 20 mg per day.
* Involvement in another experimental drug trial within the last month.
* Clinical evidence of cellulitis or infection in or around the ulcer.
* History of non-compliance to medical regimens and is not considered reliable.
* Unable to understand the study evaluations and provide a written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-03; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Tabulations of AEs (Adverse Event), review of CBC (Complete Blood Count) with differential and platelet. | CBC at initial screening and completion of dose regiment (8 weeks). AE's evaluated per protocol if and when they occur.

SECONDARY OUTCOMES:
Wound edge healing rate | Weekly
Complete Wound Closure | Weekly

CONTACTS AND LOCATIONS:
Locations (1):
- Roger Williams Medical Center, Providence, Rhode Island, United States